CLINICAL TRIAL: NCT02691546
Title: Screening for Chronic Kidney Disease (CKD) Among Older People Across Europe (SCOPE)
Acronym: SCOPE
Status: Completed | Type: Observational
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Ben-Gurion University of the Negev (Other); Erasmus Medical Center (Other); Medical University of Graz (Other); Servicio Madrileño de Salud, Madrid, Spain (Other); Institut Catala de Salut (Other Government); UNIVERSYTET MEDYCZNY W LODZI (Unknown); Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: INRCA_01_2016; Grant Agreement n. 634869 (Other Grant/Funding Number: European Commission-Horizon 2020)
Record Dates: First submitted 2016-02-20; First posted 2016-02-25 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2016-02

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Diseases; Older; Geriatric assessment; Biomarkers
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum, whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects aged 75 years or older
  Interventions: Other: blood sample collection

INTERVENTIONS:
Other: blood sample collection

SUMMARY:
The SCOPE study is an observational, multicenter, prospective cohort study aimed at evaluating a 2-year screening programme for CKD in a population of older patients, aged 75 years or more, in seven European Countries, in an attempt to investigate whether and to which extent currently available screening methods may identify older people at risk of worsening kidney function.

ELIGIBILITY:
Inclusion Criteria:

* age≥75 years
* subjects attending the outpatient services at participating institutions

Exclusion Criteria:

* ESRD or dialysis
* history of solid organ or bone marrow transplantation
* active malignancy within 24 months prior to screening or metastatic cancer
* life expectancy less than 6 months
* severe cognitive impairment (MMSE<10),
* any medical or other reason that the subject is unsuitable for the study
* subjects unwilling to provide consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: subjects with 75 years or older
Sampling Method: Non-Probability Sample
Enrollment: 2434 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Rate of estimated Glomerular Filtration Rate (eGFR) decline | 24 months
  eGFR will be calculated using the Berlin Initiative Study 1 (BIS1) equation
Incidence of End Stage Renal Disease (ESRD) | 24 months
  ESRD will be defined as eGFR<15 mL/min/1.73 m2 or dialysis

SECONDARY OUTCOMES:
Biomarkers of kidney function | Baseline and 24 months
  cystatin C, beta2-microglobulin, beta-trace protein
Genetic and epigenetic analyses | Baseline and 24 months
  circulating microRNA, telomere length in circulating leukocytes, DNA methylation, analysis of the whole genome
Incidence of CKD complications | 24 months
  anemia, hyperphosphatemia, acidosis, hypoalbuminemia, hyperparathyroidism, hyperkaliemia
Incidence of major comorbidities | 24 months
  myocardial infarction, hospitalization for unstable angina, transient ischemic attack/stroke, heart failure events, interventional cardiology events, peripheral vascular intervention, and stent thrombosis
Cardiovascular mortality | 24 months
  death resulting from acute myocardial infarction, sudden cardiac death, heart failure, stroke, CV procedures, CV hemorrhage, and other CV causes
Comprehensive geriatric assessment (CGA) | Baseline and 24 months
  Cognitive function (Mini Mental State Examination), depression (Geriatric Depression Scale), functional assessment (Basic Activity of Daily Living, Lawton Instrumental Activities of Daily Living Scale), health status (Cumulative Illness Rating Scale for Geriatrics), risk of malnutrition (Mini Nutritional Assessment), dietary intake assessment (24-h Dietary Recall), history of falls and incident falls, vision and hearing impairment, socioeconomic Status, physical Performance (Short Physical Performance Battery Test), muscle strength (Hand Grip Strength), quality of life (Euro-Qol 5D)
Healthcare resource consumption | Baseline and 24 months
  previous physician visits, use of care services, hospital admissions, laboratory tests performed

CONTACTS AND LOCATIONS:
Locations (9):
- MEDIZINISCHE UNIVERSITAT- Internal Medicine/Nephrology/Geriatric Department, Graz, Austria
- FRIEDRICH-ALEXANDER-UNIVERSITAT-Institute for Biomedicine of Aging, Erlangen, Germany
- BEN-GURION UNIVERSITY-Geriatrics Department, Beersheba, Israel
- Italy (2):
  - INRCA Research Hospital, Ancona
  - INRCA Research Hospital, Cosenza
- ERASMUS UNIVERSITAIR MEDISCH CENTRUM-Department of Internal Medicine, Rotterdam, Netherlands
- UNIVERSYTET MEDYCZNY-Department of Geriatrics, Lodz, Poland
- Spain (2):
  - INSTITUT CATALA DE LA SALUT-Internal Medicine Deparment, Barcelona
  - SERVICIO MADRILENO DE SALUD-Geriatric Department, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Freiberger E, Fabbietti P, Corsonello A, Lattanzio F, Sieber C, Tap L, Mattace-Raso F, Arnlov J, Carlsson AC, Roller-Wirnsberger R, Wirnsberger G, Moreno-Gonzalez R, Formiga F, Martinez SL, Gil P, Kostka T, Guligowska A, Yehoshua I, Melzer I, Kob R; SCOPE investigators. Short physical performance battery is not associated with falls and injurious falls in older persons: longitudinal data of the SCOPE project. Eur Geriatr Med. 2024 Jun;15(3):831-842. doi: 10.1007/s41999-024-00941-y. Epub 2024 Feb 28. PMID 38416398
- [Derived] Freiberger E, Fabbietti P, Corsonello A, Lattanzio F, Artzi-Medvedik R, Kob R, Melzer I; SCOPE consortium; Britting S. Transient versus stable nature of fear of falling over 24 months in community-older persons with falls- data of the EU SCOPE project on Kidney function. BMC Geriatr. 2022 Aug 23;22(1):698. doi: 10.1186/s12877-022-03357-0. PMID 35999522
- [Derived] Tap L, Corsonello A, Formiga F, Moreno-Gonzalez R, Arnlov J, Carlsson AC, Roller-Wirnsberger R, Wirnsberger G, Ziere G, Freiberger E, Sieber C, Kostka T, Guligowska A, Gil P, Martinez SL, Artzi-Medvedik R, Yehoshua I, Fabbietti P, Lattanzio F, Mattace-Raso F; SCOPE investigators. Is kidney function associated with cognition and mood in late life? : The Screening for CKD among Older People across Europe (SCOPE) study. BMC Geriatr. 2020 Oct 2;20(Suppl 1):297. doi: 10.1186/s12877-020-01707-4. PMID 33008359
- [Derived] Britting S, Artzi-Medvedik R, Fabbietti P, Tap L, Mattace-Raso F, Corsonello A, Lattanzio F, Arnlov J, Carlsson AC, Roller-Wirnsberger R, Wirnsberger G, Kostka T, Guligowska A, Formiga F, Moreno-Gonzalez R, Gil P, Martinez SL, Kob R, Melzer I, Freiberger E; SCOPE investigators. Kidney function and other factors and their association with falls : The screening for CKD among older people across Europe (SCOPE) study. BMC Geriatr. 2020 Oct 2;20(Suppl 1):320. doi: 10.1186/s12877-020-01698-2. PMID 33008307
- [Derived] Corsonello A, Fabbietti P, Formiga F, Moreno-Gonzalez R, Tap L, Mattace-Raso F, Roller-Wirnsberger R, Wirnsberger G, Arnlov J, Carlsson AC, Weingart C, Freiberger E, Kostka T, Guligowska A, Gil P, Martinez SL, Melzer I, Yehoshua I, Lattanzio F; SCOPE investigators. Chronic kidney disease in the context of multimorbidity patterns: the role of physical performance : The screening for CKD among older people across Europe (SCOPE) study. BMC Geriatr. 2020 Oct 2;20(Suppl 1):350. doi: 10.1186/s12877-020-01696-4. PMID 33008303
- [Derived] Corsonello A, Tap L, Roller-Wirnsberger R, Wirnsberger G, Zoccali C, Kostka T, Guligowska A, Mattace-Raso F, Gil P, Fuentes LG, Meltzer I, Yehoshua I, Formiga-Perez F, Moreno-Gonzalez R, Weingart C, Freiberger E, Arnlov J, Carlsson AC, Bustacchini S, Lattanzio F; SCOPE investigators. Design and methodology of the screening for CKD among older patients across Europe (SCOPE) study: a multicenter cohort observational study. BMC Nephrol. 2018 Oct 11;19(1):260. doi: 10.1186/s12882-018-1030-2. PMID 30309342